CLINICAL TRIAL: NCT05753124
Title: Investigation and Study of Pregnancy in Overweight or Diabetic Women and the Effect of Bariatric Surgery on Pregnancy Outcomes
Brief Title: Effect of Obesity, Diabetes and Bariatric Surgery on Pregnancy Outcomes
Status: Recruiting | Type: Observational
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 142103
Record Dates: First submitted 2022-07-04; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Pregnancy in Diabetic; Pregnancy Complications; Pregnancy Related; Bariatric Surgery Status Complicating Pregnancy
Keywords: Pregnancy; Gastric sleeve; Gastric bypass; Bariatric surgery; Birth weight; Glucose intolerance
MeSH Terms: conditions — Obesity; Pregnancy in Diabetics; Pregnancy Complications; Birth Weight; Glucose Intolerance | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal blood, urine, stool samples and vaginal swabs.
  Neonatal cord blood, urine and meconium samples.
  Maternal (after the delivery) and infant blood, urine and stool samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pregnant women with obesity/GDM/T2DM: Pregnant women with obesity/GDM/T2DM
- Pregnant women with obesity/GDM/T2DM- Controls: Pregnant women with normal BMI/ no GDM orT2DM
- Post-bariatric pregnant women: Pregnant women with previous bariatric surgery
  Interventions: Other: Observational
- Pregnant no bariatric women- Controls: There will be two control groups of women with no previous bariatric surgery:
  1. Pregnant women with booking BMI similar to the booking BMI of the post-bariatric ones and 2. Pregnant women with booking BMI similar to the pre-surgery BMI of the post-bariatric ones.

INTERVENTIONS:
Other: Observational — This is an observational study
  Groups: Post-bariatric pregnant women

SUMMARY:
The obesity epidemic is growing worldwide and in the UK this is perpetuated with a third of women classified as overweight/obese in 2020. Many of these woman are of childbearing age and go on to have high risk pregnancies which are often complicated by gestational or pre-existing (type 2 diabetes mellitus (GDM, T2DM). Bariatric surgery is the most successful treatment of sustainable weight loss and is associated with a reduction in rates of GDM, pre-eclampsia, delivery of large babies but increased risk of delivery of small babies and preterm delivery.

The aims of the study are to investigate the maternal and fetal/neonatal, biophysical and biochemical, intra-uterine environment and postnatal profile of pregnancies:

1. affected by maternal obesity and/or GDM/T2DM compared to pregnancies with normal maternal body mass index (BMI).
2. with previous maternal bariatric surgery compared to pregnancies without previous bariatric surgery but matched for maternal pre-surgery and early pregnancy BMI.

DETAILED DESCRIPTION:
This is an observational study. The investigators are planning to study pregnant women with normal BMI or overweight (BMI<30), obesity (BMI ≥30) and glucose disorders (GDM and T2DM). The investigators will also study pregnant women with previous bariatric surgery (gastric band, sleeve gastrectomy or gastric bypass) and compare them with pregnant women of similar pre-surgery and early pregnancy BMI, but no hisotry of weight loss surgery.

For all the participants and serially during pregnancy (at 12-14, 20-24, 26-28, 30-32, 35-37 weeks gestation and postnatally (at 6 weeks, 3 months, 12-24 months and 3-7 years of age), the investigators will perform the following investigations:

Maternal investigations: Demographics and medical history will be recorded, weight, height, waist to hip ratio and blood pressure will be measured, blood, urine, stool samples and vaginal swabs will be obtained, cervical length (by trans-vaginal ultrasound) will be measured and maternal echocardiography will be performed. Maternal glucose homeostasis will be assessed at 26-28 weeks of gestation, by a full oral glucose tolerance test, HOMA, home glucose monitoring and/ or continuous glucose monitoring (CGM), depending on the group the women belong to.

Fetal investigations: Fetal growth and well being will be assessed by 2D, 3D and Doppler ultrasound, fetal echocardiography will be performed.

At and following delivery: Maternal blood and urine samples and subcutaneous and omental fat (if Caesarean section is performed) will be obtained, placental tissue will be stored. Neonatal cord blood will be obtained, birthweight (percentiles), anthropometric characteristics will be measured, meconium and urine samples will be obtained and neonatal MRI (to assess body fat distribution) will be arranged.

Postnatal follow up visits for the mother and the infant (at 6 weeks, 3 months, 12-24 months, 3-7 years old) will be arranged and maternal and infant blood and urine samples will be requested and obtained.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with normal size (BMI <30)
* Pregnant women with obesity (BMI ≥30)
* Pregnant women with glucose disorders
* Pregnant women with previous bariatric surgery

Exclusion Criteria:

* Pregnant women less than 18 years of age
* Pregnant women with twins/triplets

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female and pregnant. Only looking at singleton pregnancies.
Study Population: Pregnant women with a singleton pregnancy that resulted in the delivery of a live, phenotypically normal neonate.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Birth weight (in percentiles) | At the time of birth
  Birthweight percentiles will be compared in the groups studied

SECONDARY OUTCOMES:
Reported pregnancy complications | During pregnancy and up until the birth of the baby
  Compare the percentage of women that develop pre-eclampsia or other complications in the groups studied
Reported labour outcomes | At birth
  The percentage of women who deliver by instrumental deliveries or Caesarean section, in the groups studied
Maternal and infant weight (in kg) and height (in cm) | Following the birth: 6 weeks, 3 months, 12-24 months and 3-7 years
  Weight and height will be combined to report BMI in kg/m^2, in the groups of women studied
Maternal and infant blood pressure (in mmHg) | Following the birth: 6 weeks, 3 months, 12-24 months and 3-7 years
  Compare the maternal and infant biophysical profile in the groups of women studied
Maternal and infant blood and urine samples | Following the birth: 6 weeks, 3 months, 12-24 months and 3-7 years
  Compare the maternal and infant metabolic profile in the groups of women studied

CONTACTS AND LOCATIONS:
Overall Officials: MAKRINA SAVVIDOU, MD, Principal Investigator — CHELSEA & WESTMINSTER HOSPITAL NHS FT
Locations (1):
- Chelsea & Westminster Hospital Nhs Ft, London, United Kingdom